CLINICAL TRIAL: NCT01864122
Title: Predictive Value of Coronary Heart Disease (CHD) Biomarkers for CHD Death
Acronym: WHI
Status: Completed | Type: Observational
Sponsor: Tufts University (Other)
Collaborators: Northwestern University (Other); Fred Hutchinson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 8141
Record Dates: First submitted 2013-05-03; First posted 2013-05-29 (Estimated); Last update posted 2025-05-06 (Actual); Status verified 2017-10

CONDITIONS: Cardiovascular Disease
Keywords: nutrient biomarkers; food frequency questionnaire; predictors of CVD; fatty acids; phylloquinone; dihydrophylloquinone
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The overall objective of this research proposal is to determine whether the predictive value of using plasma concentrations of selected nutrient biomarkers of food intake determined using a single plasma sample either alone or in combination are stronger, objective predictors of subsequent death from coronary heart disease (CHD) or myocardial infarct (MI) compared to selected food intake data derived from subjective, self-reported food frequency questionnaires.

DETAILED DESCRIPTION:
The overall objective is to determine whether the predictive value of plasma concentrations of selected nutrient biomarker(s) of food intake determined using a single plasma sample either alone or in combination are stronger, objective predictors of subsequent death from CHD or MI compared to selected food intake data derived from subjective, self-reported food frequency questionnaires. The nutrient biomarkers (phospholipid [PL] eicosapentaenoic acid [EPA], PL docosahexaenoic acid [DHA], PL trans fatty acids, phylloquinone, dihydrophylloquinone) and foods (fish, dark fish and tuna, vegetables, fruits, and whole grains, and unsaturated fat rich foods) targeted have previously been either directly or indirectly associated with CVD risk. We propose to test our overall objective by conducting a nested case-control study using plasma samples and food frequency data from the observational cohort of the Women's Health Initiative (WHI). Our cases (n=1200) will be selected from the subset of women who did not report dietary supplement use and who died of CHD or MI (collectively referred to as WHI CHD cases). The control subjects (n=1200) will be selected from the subset that were free of CHD or MI events and matched with cases for standard National Cholesterol Education Program (NCEP) risk factors (WHI controls). Nutrient biomarker data will be newly generated using stored specimens whereas the selected food intake data have previously been collected by the WHI investigators.

ELIGIBILITY:
Inclusion Criteria:

Cases, defined as women with centrally confirmed CHD and fatal or non-fatal myocardial infarction (MI).

Control subjects were matched on the basis of age, enrollment date, race/ethnicity and absence of CHD, MI, angina, coronary artery by-pass graft/ percutaneous transluminal coronary angioplasty, congestive heart failure, stroke or peripheral vascular disease at baseline.

Exclusion Criteria:

none

Min Age: 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Womens' Health Initiative Observational Study
Sampling Method: Non-Probability Sample
Enrollment: 2448 (Actual)
Dates: Start 2007-01; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
plasma markers of dietary intake | 4 years
  phospholipid fatty acid profiles

SECONDARY OUTCOMES:
self-reported food frequency questionnaire data analysis | 2 years
  analysis of data generated from self-reported food questionnaire, documenting types and amounts and frequency of foods consumed
phylloquinone | 4 years
  quantification of phylloquinones
dihydrophylloquinone | 4 years
  quantification of dihydrophylloquinones
desaturase indexes | 4 years
  determination of desaturase indexes
carotenoids | 4 years
  quantification of carotenoids

CONTACTS AND LOCATIONS:
Overall Officials: Alice H Lichtenstein, D.Sc., Principal Investigator — Tufts University
Locations (1):
- Tufts University, Boston, Massachusetts, United States

REFERENCES:
- [Background] Horn LV, Tian L, Neuhouser ML, Howard BV, Eaton CB, Snetselaar L, Matthan NR, Lichtenstein AH. Dietary patterns are associated with disease risk among participants in the Women's Health Initiative Observational Study. J Nutr. 2012 Feb;142(2):284-91. doi: 10.3945/jn.111.145375. Epub 2011 Dec 21. PMID 22190026
- [Background] Matthan NR, Ooi EM, Van Horn L, Neuhouser ML, Woodman R, Lichtenstein AH. Plasma phospholipid fatty acid biomarkers of dietary fat quality and endogenous metabolism predict coronary heart disease risk: a nested case-control study within the Women's Health Initiative observational study. J Am Heart Assoc. 2014 Aug 13;3(4):e000764. doi: 10.1161/JAHA.113.000764. PMID 25122663